CLINICAL TRIAL: NCT07266051
Title: Prospective Cohort Study of Neuromyelitis Optica Spectrum Disorders (NMOSD)
Acronym: NMOSD
Status: Not yet recruiting | Type: Observational
Sponsor: Xiamen Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Li Shiyong, Xiamen Traditional Chinese Medicine Hospital, Xiamen Hospital of Traditional Chinese Medicine
Other Study IDs: 2025-K065-01
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: NMOSD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MNOSD patient group: The NMOSD patient cohort consisted of adults (≥18 years) who met the 2021 Chinese diagnostic criteria, were AQP4-IgG seropositive, and provided informed consent.
  Interventions: Other: Sex hormone assay
- Healthy control group: Age- and sex-matched healthy controls (≥18 years) who provided informed consent
  Interventions: Other: Sex hormone assay

INTERVENTIONS:
Other: Sex hormone assay — This study will explore and validate the characteristics of sex hormone levels in MNMOSD
  Groups: MNOSD patient group
Other: Sex hormone assay — This study will explore the comparison of sex hormone levels between a healthy control group and MNMOSD
  Groups: Healthy control group

SUMMARY:
This study aims to characterize sex hormone alterations and their potential clinical significance in NMOSD patients from Southern China through comprehensive hormonal profiling.

DETAILED DESCRIPTION:
This study is a prospective cohort study, aiming to explore the characteristics of sex hormone levels in patients with neuromyelitis optica spectrum disorder (NMOSD). It plans to include 2,000 patients with NMOSD and 2,000 healthy controls, and conduct a 3-year follow-up. By regularly collecting data such as serum sex hormone levels, imaging, neurological function scales, and various biomarkers, the differences between the two groups will be compared and analyzed to reveal the role of sex hormones in NMOSD and their association with disease activity.

ELIGIBILITY:
Inclusion Criteria Inclusion Criteria for the NMOSD Patient Group

* Aged 18 years or older, regardless of sex
* Fulfilled the diagnostic criteria for Neuromyelitis Optica Spectrum Disorders as defined by the 2021 Chinese guidelines for the diagnosis and management of NMOSD
* Seropositive for AQP4-IgG
* Provided informed consent by the participant or their legal guardian

Inclusion Criteria for the Healthy Control Group

* Aged 18 years or older, regardless of sex
* Gender- and age-matched healthy individuals
* Provided informed consent by the participant or their legal guardian

Exclusion Criteria

* Diagnosis of other serious systemic diseases (e.g., malignancy)
* Presence of severe psychiatric disorders that would preclude compliance with study procedures and/or follow-up assessments
* History of infectious pathologies of the central nervous system
* Those with severe liver and kidney function impairment or dysfunction of other vital organs
* Patients with other conditions that do not allow participation in clinical research
* Patients allergic to gadolinium-DPTA
* Patients with other conditions that do not allow participation in clinical research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of NMOSD patients in Southern China
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-07 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Variations in Serum Sex Hormones | Baseline, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyong Li, Study Chair — Xiamen Hospital of Traditional Chinese Medicine
Locations (5):
- China (5):
  - The First Affiliated Hospital of Xiamen university, Xiamen, Fujian
  - The Second Affiliated Hospital of Xiamen Medical College, Xiamen, Fujian
  - Xiamen Hospital of Traditional Chinese Medicine, Xiamen, Fujian
  - Zhongshan Hospital (Xiamen), Fudan University, Xiamen, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian